CLINICAL TRIAL: NCT06220929
Title: The Effect of the Combination of Mecobalamin and Ceftriaxone Sodium on Liver Injury in Sepsis and Clinical Prognosis Observation
Brief Title: Mecobalamin Combined With Ceftriaxone Sodium in the Treatment of Sepsis Liver Injury
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Chun Pan, Principal investigater, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPan
Record Dates: First submitted 2024-01-13; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Sepsis; Liver Dysfunction
MeSH Terms: conditions — Sepsis; Liver Diseases | interventions — mecobalamin; Ceftriaxone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Patients were randomly divided into intervention and control groups, with both groups receiving standard treatment and care for sepsis (decided by the attending physician). On this basis, the following treatments were administered: Control group (n=20): intravenous saline drip/oral placebo tablets.
  Interventions: Drug: Saline; Drug: Placebo
- Intervention group (Experimental): Patients were randomly divided into intervention and control groups, with both groups receiving standard treatment and care for sepsis (decided by the attending physician). On this basis, the following treatments were administered: Intervention group (n=20): intravenous drip of ceftriaxone sodium 1g per dose, twice daily (continuously for 14 days), mecobalamin injection 1mg per dose, once daily (on days 1, 2, 3, 5, 7, 9, 11, 13), with a half-hour interval between medications. From day 15 to 28, take mecobalamin tablets orally, 1mg per dose, three times a day.
  Interventions: Drug: Mecobalamin; Drug: Ceftriaxone Sodium

INTERVENTIONS:
Drug: Mecobalamin — The drug Mecobalamin in the intervention group was divided into intravenous and oral formulations, with the intravenous formulation being used for the first 14 days of the experiment and the oral formulation for the second 14 days.
  Arms: Intervention group
Drug: Ceftriaxone Sodium — Ceftriaxone sodium all intravenous formulations
  Arms: Intervention group
Drug: Saline — The saline used in the control group was the same as the saline used in the experimental group to dispense the drug
  Arms: Control group
Drug: Placebo — Placebo and Mecobalamin tablets look and smell the same.
  Arms: Control group

SUMMARY:
The previous research of our research group shows that during the course of sepsis, the pyroptosis mediated by the caspase-4/GSDMD pathway in immune cells, induced by pathogens, is the main cause of immune collapse in sepsis patients. The preliminary study of this project further reveals that sepsis combined with intrahepatic cholestasis subsequently induces a rapid hepatocyte pyroptosis mediated by the Apaf-1 pyroptosome/caspase-3/GSDME signaling pathway. The interaction of these two processes triggers liver organ failure, suggesting GSDMD/GSDME as targets for the treatment of liver damage/liver failure in sepsis . Based on high-throughput drug screening and validation in in vivo and in vitro models, it was found that the combination of the old drug mecobalamin with ceftriaxone sodium, or with thiamine, used therapeutically, can block both of these cell pyroptosis pathways. Compared with corticosteroid drugs like dexamethasone and liver-protecting drugs, they have superior effects. Patients were randomly divided into intervention and control groups, with both groups receiving standard treatment and care for sepsis (decided by the attending physician). On this basis, the following treatments were administered: Control group (n=20): intravenous saline drip/oral placebo tablets; Intervention group (n=20): intravenous drip of ceftriaxone sodium 1g per dose, twice daily (continuously for 14 days), mecobalamin injection 1mg per dose, once daily (on days 1, 2, 3, 5, 7, 9, 11, 13), with a half-hour interval between medications. From day 15 to 28, take mecobalamin tablets orally, 1mg per dose, three times a day.

DETAILED DESCRIPTION:
1. Eligibility Criteria (1) Mild to moderate sepsis as defined by the △SOFA score; (2) Admission to ICU <24 hours; (3) Serum total bile acid concentration TBA ≥10μmol/L, total bilirubin concentration TBiL ≥17.1 μmol/L; (4) Patients with suspected or confirmed infection as the main cause.
2. Exclusion Criteria (1) Age >85 years or <18 years; (2) Patients contraindicated for mecobalamin treatment, allergic to ceftriaxone sodium, or other contraindications; (3) Existence of a potential disease with a life expectancy of <1 year; (4) Patients with non-infectious causes such as burns, trauma, chemical poisoning; (5) Withdrawal of life support or anticipated life-threatening condition within 48 hours; (6) History of autoimmune diseases, tumors, hepatobiliary diseases, diabetes, metabolic genetic diseases; (7) Vitamin B deficiency, malnutrition history; (8) Re-admission to ICU within one year; (9) Relatives or guardians unwilling to participate in the study; (10) Pregnancy.
3. Withdrawal Criteria (1) Adverse reactions related to mecobalamin or ceftriaxone sodium treatment; (2) Rapid progression of disease requiring treatment adjustment; (3) Other life-threatening reasons as decided by the clinician to stop the trial; (4) Patient or guardian request to withdraw from the trial.
4. Termination Criteria (1) Severe or intolerable adverse events (e.g., severe liver and kidney dysfunction), necessitating withdrawal from the trial as judged by the researchers; (2) Decision by the patient and family to withdraw from the study at any stage; (3) Discontinuation of participation in the study as deemed necessary by the attending physician based on the patient's condition.
5. Study Content 5.1 Screening Period Within 24 hours before enrollment, perform blood routine, liver and kidney function tests, and interviews. Select sputum, blood, and other fluid samples based on potential infection sites for smear and Gram staining microscopy. Concurrently conduct blood culture and drug sensitivity tests to assess the most likely pathogens causing infection. Randomly assign patients into either the placebo group or the ceftriaxone group following the principle of random controlled trials, done by a computer system (like drawing lots) at a 1:1 ratio. The process is uncontrollable by doctors or others. All trial drug packages look the same and can only be identified by a unique trial identifier. Group assignment and drug numbering are managed by a designated person. The appearance of the drug boxes for both groups is identical, and the attending physicians and patients are unaware of whether the drugs in the numbered boxes are placebo or therapeutic. The bedside nurses are responsible for administering the numbered drugs according to the plan, thus ensuring blinding of the trial participants and all research center staff to ceftriaxone, mecobalamin, or placebo.

   5.2 Intervention Period Both groups receive standard sepsis treatment and care (decided by the attending physician). Additional treatments are as follows: 1) Control group (n=20): intravenous saline drip/oral placebo tablets; 2) Mecobalamin + ceftriaxone sodium group (n=20): intravenous drip of ceftriaxone sodium 1g per dose, twice daily (for 14 consecutive days), and mecobalamin injection 1mg per dose, once daily (on days 1, 2, 3, 5, 7, 9, 11, 13), with at least a half-hour interval between medications. From day 15 to 28, take mecobalamin tablets orally, 1mg per dose, three times a day.

   5.3 Follow-up Period 5.3.1 Main Indicators (1) General data: Admission basic materials (name, gender, date of birth, height, actual weight, etc.), ICU admission details (time of joining the group, APACHEII score, SOFA score, Glasgow score, main diagnosis, medical history, etc.), pre-enrollment treatment and medication records. (2) On days 1, 3, 7, 14, and 28 or before transfer from ICU: organ failure (SOFA score), ALT, AST, total bilirubin, direct bilirubin, indirect bilirubin, bile acids, blood ammonia, coagulation function, blood gases, vasoactive drugs, kidney function, serum lactate. (3) Liver ultrasound imaging on days 1, 7, 14, or before ICU transfer.

   Note: Organ failure is measured by the Sequential Organ Failure Assessment (SOFA) score, grading the function of six organ systems based on blood pressure and vasoactive drug needs, oxygenation, platelet count, serum creatinine, and bilirubin levels, as well as the Glasgow Coma Scale score. The severity of illness is measured by the Acute Physiology and Chronic Health Evaluation (APACHE) II, ranging from 0 to 71, with higher scores indicating a higher risk of death.
6. Evaluation Indicators/Study Endpoints 6.1 Primary Observation Endpoint Improvement in liver function by 28 days or at discharge/death: Total bilirubin reduced to ≤17.1μmol/L and bile acids <10μmol/L.

   6.2 Secondary Observation Endpoints (1) 28-day mortality rate; (2) ICU and hospital stay duration; (3) Number of days without organ dysfunction in 28 days; (4) Changes in serum markers related to cell pyroptosis and tissue necrosis, such as interleukins-1β, 1α, LDH, etc.
7. Visit Arrangement and Data Collection During the Study (1) General data: Admission basic materials (name, gender, date of birth, height, actual weight, etc.), ICU admission details (time of joining the group, APACHEII score, SOFA score, Glasgow score, main diagnosis, medical history, etc.), pre-enrollment treatment and medication records. (2) On days 1, 3, 7, 14, and 28 or before transfer from ICU: organ failure (SOFA score), ALT, AST, total bilirubin, direct bilirubin, indirect bilirubin, bile acids, blood ammonia, coagulation function, blood gases, vasoactive drugs, kidney function, serum lactate. (3) Liver ultrasound imaging on days 1, 7, 14, or before ICU transfer.

ELIGIBILITY:
Inclusion Criteria:

1. Mild to moderate sepsis as defined by the △SOFA score;
2. Admission to ICU <24 hours;
3. Serum total bile acid concentration TBA ≥10μmol/L, total bilirubin concentration TBiL ≥17.1 μmol/L;
4. Patients with suspected or confirmed infection as the main cause.-

Exclusion Criteria:

1. Age >85 years or <18 years;
2. Patients contraindicated for mecobalamin treatment, allergic to ceftriaxone sodium, or other contraindications;
3. Existence of a potential disease with a life expectancy of <1 year;
4. Patients with non-infectious causes such as burns, trauma, chemical poisoning;
5. Withdrawal of life support or anticipated life-threatening condition within 48 hours;
6. History of autoimmune diseases, tumors, hepatobiliary diseases, diabetes, metabolic genetic diseases;
7. Vitamin B deficiency, malnutrition history;
8. Re-admission to ICU within one year;
9. Relatives or guardians unwilling to participate in the study;
10. Pregnancy.-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
total bilirubin | 28 days or when patient is discharged/dead
  Total bilirubin reduced to 17.1 μmol/L
bile acids | 28 days or when patient is discharged/dead
  Bile acids <10 μmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Chun Pan, ph.D, Study Director — Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lelubre C, Vincent JL. Mechanisms and treatment of organ failure in sepsis. Nat Rev Nephrol. 2018 Jul;14(7):417-427. doi: 10.1038/s41581-018-0005-7. PMID 29691495
- [Background] He XL, Chen JY, Feng YL, Song P, Wong YK, Xie LL, Wang C, Zhang Q, Bai YM, Gao P, Luo P, Liu Q, Liao FL, Li ZJ, Jiang Y, Wang JG. Single-cell RNA sequencing deciphers the mechanism of sepsis-induced liver injury and the therapeutic effects of artesunate. Acta Pharmacol Sin. 2023 Sep;44(9):1801-1814. doi: 10.1038/s41401-023-01065-y. Epub 2023 Apr 11. PMID 37041228
- [Background] Jiao C, Zhang H, Li H, Fu X, Lin Y, Cao C, Liu S, Liu Y, Li P. Caspase-3/GSDME mediated pyroptosis: A potential pathway for sepsis. Int Immunopharmacol. 2023 Nov;124(Pt B):111022. doi: 10.1016/j.intimp.2023.111022. Epub 2023 Oct 12. PMID 37837715
- [Background] Pan C, Chen L, Lu C, Zhang W, Xia JA, Sklar MC, Du B, Brochard L, Qiu H. Lung Recruitability in COVID-19-associated Acute Respiratory Distress Syndrome: A Single-Center Observational Study. Am J Respir Crit Care Med. 2020 May 15;201(10):1294-1297. doi: 10.1164/rccm.202003-0527LE. No abstract available. PMID 32200645